CLINICAL TRIAL: NCT05397431
Title: Specific Use-Results Survey of TAKHZYRO Subcutaneous Injection 300 mg Syringe for Hereditary Angioedema With Long-term Administration
Brief Title: A Survey of Lanadelumab in Participants With Hereditary Angioedema
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4004; jRCT2031220105 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lanadelumab: Participants will receive 300 milligram (mg) of Lanadelumab Subcutaneous (SC) injection once every 2 weeks.
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Lanadelumab 300 mg, subcutaneous injection every 2 weeks
  Other Names: SHP643 (TAK-743); TAKHZYRO

SUMMARY:
This study is a survey in Japan of Lanadelumab used to treat people with hereditary angioedema (HAE). The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from Lanadelumab and to check if Lanadelumab improves symptoms of HAE. During the study, participants with HAE will take Lanadelumab subcutaneous injection according to their clinic's standard practice. The study doctors will check for side effects from Lanadelumab for 12 months.

ELIGIBILITY:
Inclusion Criteria - Participants diagnosed with hereditary angioedema (HAE) and treated with Lanadelumab for the first time.

Exclusion Criteria

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced At Least One Treatment-Emergent Adverse Event (TEAE) | 12 Months
  An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product. An adverse event does not necessarily have a causal relationship with the intervention. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

SECONDARY OUTCOMES:
Number of Angioedema Attacks | 12 Months
  Number of angioedema attacks during the study will be assessed.
Angioedema Quality of life (AE-QoL) Questionnaire | 12 Months
  The AE-QoL questionnaire is a self-administered validated instrument to assess health related (HR)QoL among participants with recurrent angioedema (including HAE). The AE-QoL consists of 17 disease-specific quality-of-life items, to produce a total AE-QoL score and 4 domain scores (functioning, fatigue/mood, fear/shame, and nutrition) and each of the 17 items has a five-point response scale ranging from 1 (Never) to 5 (Very Often).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6d5657d5baac48b7